CLINICAL TRIAL: NCT01613599
Title: Prospective, Observational Safety Study of Patients With Granulomatosis With Polyangiitis (Wegener's) or Microscopic Polyangiitis Treated With Rituximab
Brief Title: An Observational Study of The Safety of MabThera/Rituxan (Rituximab) in Participants With Granulomatosis With Polyangiitis (Wegener's) or Microscopic Polyangiitis
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WA27893
Record Dates: First submitted 2012-06-04; First posted 2012-06-07 (Estimated); Results first posted 2016-08-17 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Granulomatosis With Polyangiitis; Microscopic Polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Rituximab: Participants with granulomatosis with polyangiitis (GPA) (Wegener's granulomatosis) or microscopic polyangiitis (MPA) who received rituximab as per investigator's discretion were followed for a maximum of 4 years.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Participants received rituximab at the discretion of their treating physicians.
  Other Names: Rituxan

SUMMARY:
This prospective observational study will evaluate the long-term safety of MabThera/Rituxan (rituximab) in participants with granulomatosis with polyangiitis (Wegener's) or microscopic polyangiitis. Data will be collected for a maximum of 4 years from participants initiated on MabThera/Rituxan therapy by their physician according to prescribing information.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA), according to Chapel Hill Consensus Conference Definitions for MPA and American College of Rheumatology (ACR) Criteria for the Classification of GPA
* Disease severity requiring rituximab treatment per the investigator's assessment

Exclusion Criteria:

* Prior use of rituximab (except if received within 4 weeks of screening)
* Known hypersensitivity to rituximab, to any component of the product, or to murine proteins
* Pregnant or breastfeeding women
* Diagnosis of Churg-Strauss syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with granulomatosis with polyangiitis or microscopic polyangiitis treated with MabThera/Rituxan
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-06-20 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (15):
- United States (15):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Asthma&Allergy, Baltimore, Maryland
  - Mass. General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic Rochester; Int.Med - Div. of Pul, Rochester, Minnesota
  - Weill Medical College of Cornell University; Hospital for Special Surgery, New York, New York
  - UNC- Chapel Hill, Chapel Hill, North Carolina
  - Duke Univ Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah; Division of Rheumatology, Salt Lake City, Utah

REFERENCES:
- [Derived] Merkel PA, Niles JL, Mertz LE, Lehane PB, Pordeli P, Erblang F. Long-Term Safety of Rituximab in Granulomatosis With Polyangiitis and in Microscopic Polyangiitis. Arthritis Care Res (Hoboken). 2021 Sep;73(9):1372-1378. doi: 10.1002/acr.24332. Epub 2021 Aug 13. PMID 32475029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 participants were enrolled in 15 investigational sites in United States. 3 participants out of 100 enrolled participants were not included in the analysis population as that site became unresponsive.
Groups:
- Rituximab: Participants with granulomatosis with polyangiitis (GPA) (Wegener's granulomatosis) or microscopic polyangiitis (MPA) who received rituximab as per investigator's discretion were followed for a maximum of 4.32 years.
Period: Overall Study
Arm/Group | Rituximab
Started | 97
Completed | 72
Not Completed | 25
Not completed — Death | 9
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 8
Not completed — Reason not specified | 3

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received any active dose of rituximab.
Groups:
- Rituximab: Participants with GPA (Wegener's granulomatosis) or MPA who received rituximab as per investigator's discretion were followed for a maximum of 4.32 years.
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Serious Infections
Description: A serious infection was defined as an infection that was a serious adverse event (SAE) or a non-SAE infection that required treatment with intravenous antimicrobials. A SAE was defined as any adverse event that fulfilled at least one of the following criteria: •Was fatal (results in death) •Was life-threatening •Required in-patient hospitalization or prolongation of existing hospitalization •Resulted in persistent or significant disability/incapacity •Was a congenital anomaly/birth defect •Was medically significant or required intervention to prevent one or other of the outcomes listed above. Multiple events reported in the same participant were counted multiple times in the calculation of incidence. Incidence rate is defined as events per 100 patient years.
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Number analyzed (Total Patient-years at Risk) | 338
events per 100 patient year | 7.11 [4.55 to 10.58]

2. Secondary Outcome: Percentage of Participants With a Serious Infusion-related Reaction
Description: A serious infusion-related reaction was defined as a SAE during or within 24 hours after any rituximab infusion and considered infusion related by the Principal Investigator. A SAE was defined as any adverse event that fulfilled at least one of the following criteria: •Was fatal (results in death) •Was life-threatening •Required in-patient hospitalization or prolongation of existing hospitalization •Resulted in persistent or significant disability/incapacity •Was a congenital anomaly/birth defect •Was medically significant or required intervention to prevent one or other of the outcomes listed above.
Time Frame: From the start of an infusion up to 24 hours following infusion completion (Up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 97
percentage of participants | 0

3. Secondary Outcome: Incidence Rate of Serious Cardiac Adverse Events
Description: A serious cardiac adverse event was defined as a SAE that was coded to the Medical Dictionary for Regulatory Activities (MedDRA) cardiac system organ class. A SAE was defined as any adverse event that fulfilled at least one of the following criteria: •Was fatal (results in death) •Was life-threatening •Required in-patient hospitalization or prolongation of existing hospitalization •Resulted in persistent or significant disability/incapacity •Was a congenital anomaly/birth defect •Was medically significant or required intervention to prevent one or other of the outcomes listed above. Multiple events reported in the same participant were counted multiple times in the calculation of incidence. Incidence rate is defined as events per 100 patient years.
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Number analyzed (Total Patient-years at Risk) | 338
events per 100 patient year | 5.03 [2.93 to 8.06]

4. Secondary Outcome: Percentage of Participants With Any Serious Adverse Events During or Within 24 Hours After Any Rituximab Infusion
Description: A SAE was defined as any adverse event that fulfilled at least one of the following criteria: •Was fatal (results in death) •Was life-threatening •Required in-patient hospitalization or prolongation of existing hospitalization •Resulted in persistent or significant disability/incapacity •Was a congenital anomaly/birth defect •Was medically significant or required intervention to prevent one or other of the outcomes listed above.
Time Frame: From the start of an infusion up to 24 hours following infusion completion (Up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 97
percentage of participants | 0

5. Secondary Outcome: Incidence Rate of Serious Vascular Adverse Events
Description: A serious vascular adverse event was defined as a SAE coded to the MedDRA vascular system organ class. A SAE was defined as any adverse event that fulfilled at least one of the following criteria: •Was fatal (results in death) •Was life-threatening •Required in-patient hospitalization or prolongation of existing hospitalization •Resulted in persistent or significant disability/incapacity •Was a congenital anomaly/birth defect •Was medically significant or required intervention to prevent one or other of the outcomes listed above. Multiple events reported in the same participant were counted multiple times in the calculation of incidence. Incidence rate is defined as events per 100 patient years.
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Number analyzed (Total Patient-years at Risk) | 338
events per 100 patient year | 2.37 [1.02 to 4.67]

6. Secondary Outcome: Incidence Rate of Malignancy, Excluding Non-melanoma Skin Cancer
Description: Malignancies were clinical findings of cancer and excluded non-melanoma skin cancer. Multiple events reported in the same participant were counted multiple times in the calculation of incidence. Incidence rate is defined as events per 100 patient years.
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Number analyzed (Total Patient-years at Risk) | 338
events per 100 patient year | 0.89 [0.18 to 2.60]

7. Secondary Outcome: Incidence Rate of Serious Adverse Events
Description: A SAE was defined as any adverse event that fulfilled at least one of the following criteria: •Was fatal (results in death) •Was life-threatening •Required in-patient hospitalization or prolongation of existing hospitalization •Resulted in persistent or significant disability/incapacity •Was a congenital anomaly/birth defect •Was medically significant or required intervention to prevent one or other of the outcomes listed above. Multiple events reported in the same participant were counted multiple times in the calculation of incidence. Incidence rate is defined as events per 100 patient years.
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Number analyzed (Total Patient-years at Risk) | 338
events per 100 patient year | 27.84 [22.50 to 34.07]

8. Secondary Outcome: Incidence Rate of Adverse Events With Fatal Outcomes
Description: Incidence rate is defined as events per 100 patient years.
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The safety population included all participants who received any active dose of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 97
Number analyzed (Total Patient-years at Risk) | 338
events per 100 patient year | 2.67 [1.22 to 5.06]

9. Secondary Outcome: Incidence Rate of Serious Adverse Events in Participants Who Received Re-treatment With MabThera/Rituximab
Description: as for outcome 7
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: The re-treated safety population was a subset of the safety population and included all participants who received more than one course of rituximab.
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 71
Number analyzed (Total Patient-years at Risk) | 264
events per 100 patient year | 23.90 [18.36 to 30.58]

10. Secondary Outcome: Incidence Rate of Serious Infections in Participants Who Received Re-treatment With MabThera/Rituximab
Description: as for outcome 1
Time Frame: From first dose until participant withdrawal or the date of last participant, last visit (up to 4.32 years)
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: events per 100 patient year
Units Other Than Participants: Total Patient-years at Risk
Arm/Group | Rituximab
Number analyzed (Participants) | 71
Number analyzed (Total Patient-years at Risk) | 264
events per 100 patient year | 6.07 [3.47 to 9.86]

ADVERSE EVENTS:
Time Frame: Enrollment of the first participant to time of withdrawal or last participant visit (Up to 4.32 years)
Arm/Group | Rituximab
All-Cause Mortality (participants affected / at risk) | 9/97
Serious Adverse Events (participants affected / at risk) | 38/97
Other Adverse Events (participants affected / at risk) | 5/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=97)
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Staphylococcal bacteraemia (Infections and infestations) | 2
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia legionella (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothroax (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Deep vein thrombosis (Vascular disorders) | 5
Orthostatic hypotension (Vascular disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Death (General disorders) | 4
Chest pain (General disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Renal transplant (Surgical and medical procedures) | 1
Atrial tachycardia (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=97)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.